CLINICAL TRIAL: NCT04290767
Title: Evaluation of the Cerebral Microcirculation by Non-invasive Brain Ultrasound With Enhanced Microbubbles Contrast Injection in Shock Status.
Brief Title: Brain Ultrasound With Contrast Microbubbles Injection in Shock Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Duc Nam Nguyen, Clinical Professor, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B.U.N. 143201421588
Record Dates: First submitted 2020-02-12; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Shock; Microcirculation
Keywords: Shock; Brain microcirculattion; Enhanced-contrast brain ultrasound; Sulphur hexafluoride microbubbles contrast Sonovue
MeSH Terms: conditions — Shock

STUDY DESIGN:
Intervention Model Description: Cohort study in a single center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonovue (Other): ICU patients with acute shock status (septic or non-septic) who are eligible for enhanced-contrast brain ultrasound with sulphur hexafluoride microbubbles contrast (Sonovue, BRACCO, Milan, Italy) examination.
  Interventions: Diagnostic Test: Sulphur hexafluoride microbubbles SONOVUE (BRACCO, Milan, Italy)

INTERVENTIONS:
Diagnostic Test: Sulphur hexafluoride microbubbles SONOVUE (BRACCO, Milan, Italy) — Enhanced-contrast brain ultrasound with intravenously sulphur hexafluoride microbubbles SONOVUE (BRACCO, Milan, Italy) injection and using the time-intensity curve profile to evaluate brain microcirculation.

SUMMARY:
Alterations in the brain microcirculation may be involved in patients with shock. For a three-day period, we investigate the brain microcirculation using contrast-enhanced ultrasound with microbubble injection in patients with septic and non-septic shock.Ultrasound examination is performed daily to estimate global cerebral blood flow, and to evaluate the brain microcirculation, using variables of the time-intensity brain perfusion curve, after sulphur hexafluoride microbubble Sonovue injection.

DETAILED DESCRIPTION:
Non-invasive brain ultrasound with transcranial echo-color doppler (IE 33, Philips Medical System, the Netherlands) is performed in three steps to 1) evaluate the global cerebral blood volume, 2) to estimate the presence or absence of cerebral autoregulation, and 3) to qualitatively evaluate the cerebral perfusion and microcirculation by enhanced microbubbles contrast injection (CEUS). Brain ultrasound is performed in the first 48 hours after hemodynamic stabilization (MAP > 65mm Hg, normotherm) and respiratory parameters stabilization (PaCO2 between 35-45mmHg and the PaO2/FiO2 > 200) after ICU admission. The second and third examination is performed in the next 48-72 hours before sedation withdrawal to limit the effect of change of cerebral hemodynamics.

Before performing brain ultrasound, echocardiography (IE 33, Philips medical System, the Netherlands) is performed to evaluate left ventricular ejection fraction and cardiac output (L/min).

First, the global cerebral blood volume (L/min) is evaluated as the sum of flow volumes of the internal carotid (ICA) and vertebral arteries (VA) extracranial arteries of both sides. The internal carotid artery (ICA) is examined with a 7-MHz linear array transducer with the head of the patient slightly titled upward, in midline position. The site of measurement is approximately 1.5cm below the carotid bulb in the in the common carotid artery (CCA) during expansion and 1.5cm away from the bifurcation in ICA. In the presence of atheromatous calcifications plaques, ICA doppler measurement is performed outside and before the plaques. The B-mode bidimensional is magnified to achieve a higher resolution and details. The internal diameter of the vessel is measured at the exact site of the pulse doppler velocity measurement ample volume, between both endothelial layers, perpendicular of the course of the vessel. The diameter of the vertebral artery is examined and magnified in B-mode. The transducer is positioned along the CCA, shiftily laterally and angled until the intertransverse segment of the VA is seen and the doppler velocity is measured at the C4-C5 transverse area along the common carotid artery exactly at the same place of diameter measurement. The following measurements of flow velocities are taken in each artery: Peak systolic and end-diastolic velocity, time-averaged velocity (TAV), Pulsatility Index (PI). Flow volume (Q) of each artery is determined as Q = TAV x Area ((diameter of the artery /2)² x PI).

Transcranial echo-color doppler is performed via temporal windows and the Pulsatility Index (PI) and the mean flow velocities (cm/sec) are measured of MCA, at both sides are recorded. Cerebrovascular resistance index as defined as the ration MAP/Mean Flow velocity of MCA (mmHg/cm per second).

Second, after measuring the global cerebral blood volume, the presence or absence of cerebral autoregulation (CA) is tested with the Transient hyperemic response (THR) by measuring the velocity of the media cerebral artery (MCA) the following an ipsilateral common carotid compression during 8 seconds. THR is defined as the F3/F1 ratio F1 as the MCA velocity before compression and F3 is the second MCA velocity after compression test). THR test is valid when onset of compression results a sudden and maximal decrease in MCA blood velocity and remains stable during compression.

Third, after testing the THR, the brain regional microcirculation is evaluated by the microbubbles contrast injection SONOVUE (Italy) following the European guidelines recommendation for contrast microbubbles enhanced ultrasound. The brain parenchyma is insonated via the temporal bone windows at the depth of 10cm with the ultrasound S5 multifrequency transducer 2-5 MHz probe. After optimizing the acoustic bone window, SONOVUE is injected intravenously as a bolus 2.4ml followed by 10ml saline flushed. The contralateral brain is evaluated 5 minutes after the first injection of SONOVUE to allow a complete evacuation of contrast microbubbles.

All real-time CEUS images were stored digitally on the hard disk as DICOM (Digital Image Communications in Medicine) images. Offline analysis used the QLAB 10 quantification software (Philips Medical System, the Netherlands) to convert brain perfusion images into time-intensity curves (TIC) corresponding to the five different regions of interest (ROI) of brain parenchyma: anterior and posterior thalamus, lentiform nucleus, parieto-temporal and posterior white matter. Four variables were extracted from these TIC curves to qualitatively evaluate the brain microcirculation: peak intensity in dB (PI), time to peak intensity in seconds (TTP), mean transit time in seconds (MTT), and area under the curve in dB/seconds (AUC) .

ELIGIBILITY:
Inclusion Criteria:

* Septic shock criteria: refractory arterial hypotension or hypoperfusion abnormalities after fluid resuscitation with serum lactate > 4mmmol/dl, oliguria and mental status alteration or delirium.
* Cardiogenic shock is defined as refractory shock associated with oliguria and mental status alteration following acute myocardial infarction or post-cardiac surgery.

Exclusion Criteria:

* Younger than 18 years old
* Pregnancy
* Diabetes
* Acute or chronic neurological disorder: epileptics, stroke, bleeding, trauma, post-neurosurgery, post- cardiac arrest, tumor, meningitis.
* Severe dementia, psychiatric or neuromuscular disability
* Acute coronary syndrome within one previous week
* Respiratory distress ARDS with arterial oxygenation less than 70mm Hg or the FiO2 / PaO2 ratio < 200
* Advanced liver cirrhosis
* Terminal renal failure with hemodialysis and high serum uremia.> 200.
* Drug intoxications. Alcohol withdrawal.
* Advanced malign diseases
* Allergy to the microbubble contrast product Sonovue ®
* Insufficient echogenicity of bilateral temporal window to ultrasound and incomplete insonation of the intracerebral arteries
* Significant intracerebral and extracerebral arteries stenosis or severe atheromatous calcifications.
* Vertebral artery hypoplasia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative evaluation of the brain microcirculation using Sonovue injection: Mean transit time (seconds) of the time intensity curve - Mean change from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  Ultrasound examination is performed daily to evaluate the brain microcirculation, using variables of the time-intensity brain perfusion curve, after Sonovue microbubble injection. We hypothesize that the mean transit time (seconds) of this curve is early prolonged in ICU non-survivors.
Qualitative evaluation of the brain microcirculation using Sonovue injection: Peak Intensity (dB) of the time intensity curve - Mean change from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  Ultrasound examination is performed daily to evaluate the brain microcirculation, using variables of the time-intensity brain perfusion curve, after Sonovue microbubble injection. We hypothesize that the peak intensity (dB) of this curve is early reduced in ICU non-survivors.
Qualitative evaluation of the brain microcirculation using Sonovue injection: Are under the curve (percentage) of the time intensity curve - Mean change from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  Ultrasound examination is performed daily to evaluate the brain microcirculation, using variables of the time-intensity brain perfusion curve, after Sonovue microbubble injection. We hypothesize that the area under the curve (percentage) of this curve is early reduced in ICU non-survivors.
Testing daily cerebral autoregulation: Transient Hyperemic response test - Absence or presence from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  The presence or absence of cerebral autoregulation is assessed using the transient hyperemic response (THR) test, which measures the change in flow velocity in the MCA following a mild 5-second compression of the ipsilateral common carotid artery (CCA) using brain ultrasound. Cerebral autoregulation is considered absent if the flow velocity in the MCA after the compression of the ipsilateral CCA is released do not increase by more than 10% compared to the value prior to compression.
  We hypothesize that cerebral autoregulation is absent in ICU non-survivors.
Qualitative evaluation of the brain microcirculation: Mean velocity of the middle cerebral artery (cm/second) - Mean change from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  Brain ultrasound is daily performed to measure the mean velocity of both middle cerebral arteries. We hypothesize that these velocities remain unchanged or even increased in ICU non-survivors.

SECONDARY OUTCOMES:
Qualitative evaluation of the brain microcirculation: Cardiac output (L/minute) - Mean change from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  Daily transthoracic echocardiography is performed to measure the aortic velocity time integral (cm) to estimate cardiac output.
  We hypothesize that cardiac output is unchanged or even increased in ICU non-survivors.
Qualitative evaluation of the brain microcirculation: Global cerebral blood flow (L/minute) - Mean change from baseline | Comparison to baseline (24 hours after ICU admission) to the second (48 hours) and third timepoints (72 or 96 hours)
  Daily duplex echo-color of the carotids and vertebral arteries is performed to estimate global cerebral blood flow (L/minute) - Mean change from baseline.
  We hypothesize that global cerebral blood flow is unchanged or even increased in ICU non-survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Duc Nam Nguyen, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piscaglia F, Nolsoe C, Dietrich CF, Cosgrove DO, Gilja OH, Bachmann Nielsen M, Albrecht T, Barozzi L, Bertolotto M, Catalano O, Claudon M, Clevert DA, Correas JM, D'Onofrio M, Drudi FM, Eyding J, Giovannini M, Hocke M, Ignee A, Jung EM, Klauser AS, Lassau N, Leen E, Mathis G, Saftoiu A, Seidel G, Sidhu PS, ter Haar G, Timmerman D, Weskott HP. The EFSUMB Guidelines and Recommendations on the Clinical Practice of Contrast Enhanced Ultrasound (CEUS): update 2011 on non-hepatic applications. Ultraschall Med. 2012 Feb;33(1):33-59. doi: 10.1055/s-0031-1281676. Epub 2011 Aug 26. No abstract available. PMID 21874631
- [Background] Powers J, Averkiou M, Bruce M. Principles of cerebral ultrasound contrast imaging. Cerebrovasc Dis. 2009;27 Suppl 2:14-24. doi: 10.1159/000203123. Epub 2009 Apr 16. PMID 19372657
- [Background] Seidel G, Meairs S. Ultrasound contrast agents in ischemic stroke. Cerebrovasc Dis. 2009;27 Suppl 2:25-39. doi: 10.1159/000203124. Epub 2009 Apr 16. PMID 19372658
- [Background] Wiesmann M, Seidel G. Ultrasound perfusion imaging of the human brain. Stroke. 2000 Oct;31(10):2421-5. doi: 10.1161/01.str.31.10.2421. PMID 11022074